CLINICAL TRIAL: NCT01954394
Title: Open-Label Extension Study of EFC12492, R727-CL-1112, EFC12732 and LTS11717 Studies to Assess the Long-Term Safety and Efficacy of Alirocumab in Patients With Heterozygous Familial Hypercholesterolemia
Brief Title: Open Label Study of Long Term Safety Evaluation of Alirocumab
Acronym: ODYSSEY OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS13463; 2013-002572-40 (EudraCT Number); U1111-1143-3810 (Other: UTN)
Record Dates: First submitted 2013-09-16; First posted 2013-10-01 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alirocumab 75 or 150 mg Q2W (Experimental): Alirocumab 75 mg or 150 mg every 2 weeks (Q2W) added to stable lipid-modifying therapy (LMT) for up to 168 additional weeks (or until the product was commercially available) in participants who completed the parent studies EFC12492, R727-CL-1112, EFC12732 and LTS11717.
  Interventions: Drug: Alirocumab; Drug: Lipid-Modifying Therapy (LMT)

INTERVENTIONS:
Drug: Alirocumab — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with a pre-filled syringe.
  Other Names: SAR236553; REGN727; Praluent
Drug: Lipid-Modifying Therapy (LMT) — Statin (rosuvastatin, simvastatin or atorvastatin) at stable dose with or without other LMT as clinically indicated.

SUMMARY:
Primary Objective:

To assess the long-term safety of alirocumab (SAR236553/REGN727) when added to lipid-lowering therapy in participants with heterozygous familial hypercholesterolemia (heFH) who had completed EFC12492 (NCT01623115), R727-CL-1112 (NCT01709500), EFC12732 (NCT01617655) and LTS11717 (NCT01507831).

Secondary Objectives:

* To evaluate the long-term efficacy of alirocumab on lipid parameters.
* To evaluate the long-term immunogenicity of alirocumab.

DETAILED DESCRIPTION:
The maximum study duration will be 176 weeks per participant.

ELIGIBILITY:
Inclusion criteria:

Participants with heFH who had completed one of the four parent studies (EFC12492, R727-CL-1112, EFC12732 and LTS11717).

Exclusion criteria:

Significant protocol deviation in the parent study; Any permanent treatment discontinuation from the parent study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 986 (Actual)
Dates: Start 2013-12-17; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (177):
- United States (44):
  - Investigational Site Number 840321, Huntsville, Alabama
  - Investigational Site Number 840341, Tempe, Arizona
  - Investigational Site Number 840334, Bell Gardens, California
  - Investigational Site Number 840319, Fountain Valley, California
  - Investigational Site Number 840336, Los Angeles, California
  - Investigational Site Number 840339, Mission Viejo, California
  - Investigational Site Number 840337, Newport Beach, California
  - Investigational Site Number 840306, Golden, Colorado
  - Investigational Site Number 840328, Washington D.C., District of Columbia
  - Investigational Site Number 840344, Atlantis, Florida
  - Investigational Site Number 840353, Clearwater, Florida
  - Investigational Site Number 840318, Fort Lauderdale, Florida
  - Investigational Site Number 840327, Jacksonville, Florida
  - Investigational Site Number 840309, Miami, Florida
  - Investigational Site Number 840351, Sarasota, Florida
  - Investigational Site Number 840315, Evanston, Illinois
  - Investigational Site Number 840305, Oakbrook Terrace, Illinois
  - Investigational Site Number 840333, Iowa City, Iowa
  - Investigational Site Number 840329, Kansas City, Kansas
  - Investigational Site Number 840345, Auburn, Maine
  - Investigational Site Number 840338, Biddeford, Maine
  - Investigational Site Number 840322, Boston, Massachusetts
  - Investigational Site Number 840346, Framingham, Massachusetts
  - Investigational Site Number 840317, St Louis, Missouri
  - Investigational Site Number 840349, St Louis, Missouri
  - Investigational Site Number 840314, Morristown, New Jersey
  - Investigational Site Number 840316, New York, New York
  - Investigational Site Number 840324, Poughkeepsie, New York
  - Investigational Site Number 840303, Charlotte, North Carolina
  - Investigational Site Number 840320, Durham, North Carolina
  - Investigational Site Number 840348, Raleigh, North Carolina
  - Investigational Site Number 840340, Cincinnati, Ohio
  - Investigational Site Number 840302, Marion, Ohio
  - Investigational Site Number 840330, Portland, Oregon
  - Investigational Site Number 840352, Beaver, Pennsylvania
  - Investigational Site Number 840308, Philadelphia, Pennsylvania
  - Investigational Site Number 840342, Scranton, Pennsylvania
  - Investigational Site Number 840304, Summerville, South Carolina
  - Investigational Site Number 840311, Dallas, Texas
  - Investigational Site Number 840312, Dallas, Texas
  - Investigational Site Number 840301, Fort Worth, Texas
  - Investigational Site Number 840343, Bountiful, Utah
  - Investigational Site Number 840354, Chesapeake, Virginia
  - Investigational Site Number 840350, Spokane, Washington
- Argentina (2):
  - Investigational Site Number 032302, Caba
  - Investigational Site Number 032301, Coronel Suárez
- Austria (3):
  - Investigational Site Number 040302, Graz
  - Investigational Site Number 040303, Sankt Stefan
  - Investigational Site Number 040301, Vienna
- Investigational Site Number 056301, Natoye, Belgium
- Bulgaria (2):
  - Investigational Site Number 100302, Sofia
  - Investigational Site Number 100301, Sofia
- Canada (6):
  - Investigational Site Number 124303, Chicoutimi
  - Investigational Site Number 124302, Montreal
  - Investigational Site Number 124301, Québec
  - Investigational Site Number 124306, Sherbrooke
  - Investigational Site Number 124305, Toronto
  - Investigational Site Number 124304, Victoria
- Czechia (8):
  - Investigational Site Number 203307, Hradec Králové
  - Investigational Site Number 203305, Prague
  - Investigational Site Number 203301, Prague
  - Investigational Site Number 203303, Prague
  - Investigational Site Number 203306, Praha 5 - Motol
  - Investigational Site Number 203309, Trutnov
  - Investigational Site Number 203304, Uherské Hradiště
  - Investigational Site Number 203302, Zlín
- Denmark (5):
  - Investigational Site Number 208301, Aalborg
  - Investigational Site Number 208306, Aarhus
  - Investigational Site Number 208302, Esbjerg
  - Investigational Site Number 208303, Roskilde
  - Investigational Site Number 208304, Svendborg
- Finland (3):
  - Investigational Site Number 246302, Joensuu
  - Investigational Site Number 246301, Kokkola
  - Investigational Site Number 246304, Vantaa
- France (6):
  - Investigational Site Number 250303, Dijon
  - Investigational Site Number 250304, Lille
  - Investigational Site Number 250302, Nantes
  - Investigational Site Number 250301, Paris
  - Investigational Site Number 250305, Pessac
  - Investigational Site Number 250306, Rennes
- Germany (5):
  - Investigational Site Number 276302, Berlin
  - Investigational Site Number 276305, Frankfurt A.M.
  - Investigational Site Number 276306, Leipzig
  - Investigational Site Number 276301, Magdeburg
  - Investigational Site Number 276307, Witten
- Investigational Site Number 348301, Baja, Hungary
- Israel (4):
  - Investigational Site Number 376302, Holon
  - Investigational Site Number 376304, Jerusalem
  - Investigational Site Number 376303, Safed
  - Investigational Site Number 376301, Tel Litwinsky
- Italy (4):
  - Investigational Site Number 380302, Chieti
  - Investigational Site Number 380304, Milan
  - Investigational Site Number 380303, Napoli
  - Investigational Site Number 380301, Palermo
- Investigational Site Number 484301, México, Mexico
- Netherlands (20):
  - Investigational Site Number 528317, Alkmaar
  - Investigational Site Number 528301, Amsterdam-Zuidoost
  - Investigational Site Number 528320, Apeldoorn
  - Investigational Site Number 528309, Delfzijl
  - Investigational Site Number 528313, Eindhoven
  - Investigational Site Number 528319, Enschede
  - Investigational Site Number 528322, Goes
  - Investigational Site Number 528325, Groningen
  - Investigational Site Number 528302, Groningen
  - Investigational Site Number 528324, Hoogeveen
  - Investigational Site Number 528318, Hoorn
  - Investigational Site Number 528305, Leiden
  - Investigational Site Number 528311, Maastricht
  - Investigational Site Number 528312, Nijmegen
  - Investigational Site Number 528315, Rotterdam
  - Investigational Site Number 528326, Rotterdam
  - Investigational Site Number 528303, Utrecht
  - Investigational Site Number 528323, Utrecht
  - Investigational Site Number 528321, Venlo
  - Investigational Site Number 528316, Waalwijk
- Norway (3):
  - Investigational Site Number 578301, Bodø
  - Investigational Site Number 578305, Oslo
  - Investigational Site Number 578304, Oslo
- Portugal (2):
  - Investigational Site Number 620302, Funchal
  - Investigational Site Number 620301, Lisbon
- Investigational Site Number 642302, Timișoara, Romania
- Russia (9):
  - Investigational Site Number 643304, Arkhangelsk
  - Investigational Site Number 643303, Kazan'
  - Investigational Site Number 643302, Moscow
  - Investigational Site Number 643308, Moscow
  - Investigational Site Number 643305, Moscow
  - Investigational Site Number 643310, Novosibirsk
  - Investigational Site Number 643301, Saint Petersburg
  - Investigational Site Number 643306, Saint Petersburg
  - Investigational Site Number 643312, Saint Petersburg
- South Africa (14):
  - Investigational Site Number 710311, Bellville
  - Investigational Site Number 710307, Bloemfontein
  - Investigational Site Number 710306, Cape Town
  - Investigational Site Number 710302, Cape Town
  - Investigational Site Number 710309, Centurion
  - Investigational Site Number 710312, Parktown
  - Investigational Site Number 710304, Parow
  - Investigational Site Number 710313, Pretoria
  - Investigational Site Number 710303, Pretoria
  - Investigational Site Number 710305, Pretoria
  - Investigational Site Number 710314, Pretoria
  - Investigational Site Number 710315, Roodepoort
  - Investigational Site Number 710310, Somerset West
  - Investigational Site Number 710308, Witbank
- Spain (15):
  - Investigational Site Number 724303, A Coruña
  - Investigational Site Number 724308, Barcelona
  - Investigational Site Number 724306, Córdoba
  - Investigational Site Number 724312, Granada
  - Investigational Site Number 724307, L'Hospitalet de Llobregat
  - Investigational Site Number 724301, Madrid
  - Investigational Site Number 724309, Madrid
  - Investigational Site Number 724305, Madrid
  - Investigational Site Number 724311, Madrid
  - Investigational Site Number 724314, Málaga
  - Investigational Site Number 724315, Quart de Poblet
  - Investigational Site Number 724310, Sabadell
  - Investigational Site Number 724313, Seville
  - Investigational Site Number 724304, Tarragona
  - Investigational Site Number 724302, Zaragoza
- Sweden (3):
  - Investigational Site Number 752302, Gothenburg
  - Investigational Site Number 752301, Stockholm
  - Investigational Site Number 752304, Stockholm
- United Kingdom (15):
  - Investigational Site Number 826318, Birmingham
  - Investigational Site Number 826304, Brighton
  - Investigational Site Number 826301, Bristol
  - Investigational Site Number 826311, Cambridge
  - Investigational Site Number 826310, Cardiff
  - Investigational Site Number 826302, Dundee
  - Investigational Site Number 826317, Liverpool
  - Investigational Site Number 826306, Liverpool
  - Investigational Site Number 826312, Manchester
  - Investigational Site Number 826303, Manchester
  - Investigational Site Number 826305, Middlesex
  - Investigational Site Number 826313, Newcastle upon Tyne
  - Investigational Site Number 826309, Reading
  - Investigational Site Number 826315, West Bromwich
  - Investigational Site Number 826316, West Bromwich

REFERENCES:
- [Derived] Dufour R, Hovingh GK, Guyton JR, Langslet G, Baccara-Dinet MT, Din-Bell C, Manvelian G, Farnier M. Individualized low-density lipoprotein cholesterol reduction with alirocumab titration strategy in heterozygous familial hypercholesterolemia: Results from an open-label extension of the ODYSSEY LONG TERM trial. J Clin Lipidol. 2019 Jan-Feb;13(1):138-147. doi: 10.1016/j.jacl.2018.11.007. Epub 2018 Nov 30. PMID 30591415
- [Derived] Farnier M, Hovingh GK, Langslet G, Dufour R, Baccara-Dinet MT, Din-Bell C, Manvelian G, Guyton JR. Long-term safety and efficacy of alirocumab in patients with heterozygous familial hypercholesterolemia: An open-label extension of the ODYSSEY program. Atherosclerosis. 2018 Nov;278:307-314. doi: 10.1016/j.atherosclerosis.2018.08.036. Epub 2018 Sep 1. PMID 30293878
- [Derived] Hovingh GK, Guyton JR, Langslet G, Dufour R, Baccara-Dinet MT, Din-Bell C, Manvelian G, Farnier M. Alirocumab dosing patterns during 40 months of open-label treatment in patients with heterozygous familial hypercholesterolemia. J Clin Lipidol. 2018 Nov-Dec;12(6):1463-1470. doi: 10.1016/j.jacl.2018.08.011. Epub 2018 Aug 30. PMID 30287210

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 177 centers in 24 countries. Overall, 986 participants who completed study EFC12492 (NCT01623115), R727-CL-1112 (NCT01709500), EFC12732 (NCT01617655) and LTS11717 (NCT01507831) were enrolled between December 2013 and December 2014.
Pre-assignment Details: The Day 1 visit of this study was: the end of treatment visit of the 78-week treatment period for participants who completed EFC12492, R727-CL-1112 and EFC12732; and the end of study visit i.e. 8 weeks after completion of the 78-week treatment period for participants who completed LTS11717.
Groups:
- Placebo to Alirocumab 75 or 150 mg Q2W: Alirocumab 75 mg or 150 mg subcutaneous (SC) injection every 2 weeks (Q2W) added to stable lipid-modifying therapy (LMT) for up to 168 weeks in participants who received placebo in the parent studies. Participants from parent study EFC12732 (NCT01617655) started with alirocumab 150 mg Q2W and participants from parent studies EFC12492 (NCT01623115), R727-CL-1112 (NCT01709500) and LTS11717 (NCT01507831) started with alirocumab 75 mg Q2W. Alirocumab doses could be either up-titrated from 75 to 150 mg Q2W or down-titrated from 150 to 75 mg Q2W from Week 12 or maintained according to the investigator judgement and low-density lipoprotein cholesterol (LDL-C) values.
- Alirocumab to Alirocumab 75 or 150 mg Q2W: Alirocumab 75 mg or 150 mg SC injection Q2W added to stable LMT for up to 168 additional weeks in participants who received Alirocumab in the parent studies. Participants from parent study EFC12732 (NCT01617655) started with alirocumab 150 mg Q2W and participants from parent studies EFC12492 (NCT01623115), R727-CL-1112 (NCT01709500) and LTS11717 (NCT01507831) started with alirocumab 75 mg Q2W. Alirocumab doses could be either up-titrated from 75 to 150 mg Q2W or down-titrated from 150 to 75 mg Q2W from Week 12 or maintained according to the investigator judgement and LDL-C values.
Period: Overall Study
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W
Started | 331 (Enrolled) | 655 (Enrolled)
Treated | 330 (Safety population) | 655 (Safety population)
Completed | 301 | 598
Not Completed | 30 | 57
Not completed — Enrolled but not treated | 1 | 0
Not completed — Adverse Event | 10 | 23
Not completed — Poor compliance to protocol | 7 | 7
Not completed — Participant Moved | 0 | 4
Not completed — Related to Study Drug administration | 2 | 2
Not completed — Other than specified above | 10 | 21

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose or part of a dose of alirocumab in this study. Participant who was not treated, was not included in any analysis.
Groups:
- Placebo to Alirocumab 75 or 150 mg Q2W: Alirocumab 75 mg or 150 mg SC injection Q2W added to stable LMT for up to 168 weeks in participants who received placebo in the parent studies. Participants from parent study EFC12732 (NCT01617655) started with alirocumab 150 mg Q2W and participants from parent studies EFC12492 (NCT01623115), R727-CL-1112 (NCT01709500) and LTS11717 (NCT01507831) started with alirocumab 75 mg Q2W. Alirocumab doses could be either up-titrated from 75 to 150 mg Q2W or down-titrated from 150 to 75 mg Q2W from Week 12 or maintained according to the investigator judgement and LDL-C values.
- Total: Total of all reporting groups
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Total
Number analyzed (Participants) | 330 | 655 | 985
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (11.4) | 54.1 (12.1) | 54.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 287 | 435
  Male | 182 | 368 | 550
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 27 | 39
  Not Hispanic or Latino | 317 | 623 | 940
  Unknown or Not Reported | 1 | 5 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 310 | 628 | 938
  Black or African American | 2 | 2 | 4
  Asian | 2 | 6 | 8
  American Indian or Alaska Native | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 4 | 7 | 11
  White/Black or African American | 6 | 5 | 11
  White/Asian | 2 | 5 | 7
  White/American Indian or Alaska Native | 1 | 0 | 1
  Black or African American/Asian | 1 | 0 | 1
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C in mg/dL from Friedewald formula (LDL-C = Total cholesterol - High-density lipoprotein cholesterol - [Triglyceride/5]). This parameter was evaluated at the baseline in the parent study (EFC12492, R727-CL-1112, EFC12732 or LTS11717).
  mg/dL | 148.8 (48.8) | 153.5 (55.3) | 152.0 (53.2)
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] — This parameter was evaluated at the baseline in the parent study (EFC12492, R727-CL-1112, EFC12732 or LTS11717).
  mmol/L | 3.854 (1.265) | 3.977 (1.432) | 3.936 (1.379)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Adverse Events (AEs)
Description: Reported AEs are treatment-emergent AEs that is AEs that developed/worsened during the 'treatment-emergent period' (the time from the first dose of alirocumab in this study up to the last dose of alirocumab received in this study +70 days). Clinically significant lab and vital sign abnormalities were to be reported as AEs.
Time Frame: Up to 10 weeks after last study drug administration (maximum of 176 weeks)
Population: All enrolled participants who received at least one dose or part of a dose of alirocumab in this study.
Measure: Number; unit: percentage of participants
Groups:
- Alirocumab: All Participants: All participants who received alirocumab/placebo in the parent studies and received alirocumab 75 mg or 150 mg SC injection Q2W added to stable LMT for up to 168 additional weeks in this study.
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 330 | 655 | 985
percentage of participants
  Any AE | 83.9 | 87.3 | 86.2
  Any Serious AE | 20.6 | 22.0 | 21.5
  Any AE leading to treatment discontinuation | 3.0 | 3.5 | 3.4

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Weeks 8, 24, 48, 72, 96, 120, 144 and 168
Description: Baseline here corresponds to the baseline in the parent study (EFC12492, R727-CL-1112, EFC12732 or LTS11717). Post-baseline on-treatment data was obtained from Week 8 onwards up to Week 168 in this study.
Time Frame: Parent Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, and 168
Population: Modified ITT (mITT) population: all enrolled and treated participants with 1 baseline (from parent study) and at least 1 post-baseline calculated LDL-C value on-treatment. "Number analyzed" = participants evaluable at specified time-points. This number decreased significantly with visit because of the possibility to switch to commercial alirocumab.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percent change
  Week 8: number analyzed (Participants) | 306 | 611 | 917
  Week 8 | -44.9 (25.9) | -43.8 (28.7) | -44.2 (27.8)
  Week 24: number analyzed (Participants) | 305 | 621 | 926
  Week 24 | -46.9 (27.5) | -46.9 (29.3) | -46.9 (28.7)
  Week 48: number analyzed (Participants) | 309 | 609 | 918
  Week 48 | -45.6 (28.0) | -47.5 (28.8) | -46.9 (28.6)
  Week 72: number analyzed (Participants) | 293 | 594 | 887
  Week 72 | -47.7 (23.5) | -47.3 (28.4) | -47.4 (26.8)
  Week 96: number analyzed (Participants) | 236 | 475 | 711
  Week 96 | -47.4 (23.8) | -48.2 (28.2) | -47.9 (26.8)
  Week 120: number analyzed (Participants) | 188 | 352 | 540
  Week 120 | -47.4 (24.0) | -46.6 (31.1) | -46.8 (28.8)
  Week 144: number analyzed (Participants) | 69 | 129 | 198
  Week 144 | -46.5 (25.8) | -49.6 (24.6) | -48.5 (25.0)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | -43.6 (13.4) | -52.2 (20.7) | -48.8 (17.8)

3. Secondary Outcome: Absolute Change From Baseline in Calculated LDL-C (mg/dL) at Weeks 8, 24, 48, 72, 96, 120, 144 and 168
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, and 168
Population: mITT population. Here, "Number analyzed" signifies participants evaluable at specified time-points. This number decreased significantly with visit because of the possibility to switch to commercial alirocumab.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
mg/dL
  Week 8: number analyzed (Participants) | 306 | 611 | 917
  Week 8 | -66.8 (45.6) | -67.1 (49.2) | -67.0 (48.0)
  Week 24: number analyzed (Participants) | 305 | 621 | 926
  Week 24 | -70.3 (49.5) | -72.7 (52.4) | -71.9 (51.4)
  Week 48: number analyzed (Participants) | 309 | 609 | 918
  Week 48 | -67.8 (49.7) | -73.9 (54.3) | -71.9 (52.8)
  Week 72: number analyzed (Participants) | 293 | 594 | 887
  Week 72 | -71.2 (44.5) | -74.9 (54.5) | -73.7 (51.4)
  Week 96: number analyzed (Participants) | 236 | 475 | 711
  Week 96 | -70.2 (45.9) | -75.9 (55.0) | -74.0 (52.2)
  Week 120: number analyzed (Participants) | 188 | 352 | 540
  Week 120 | -72.3 (45.6) | -75.2 (59.7) | -74.2 (55.2)
  Week 144: number analyzed (Participants) | 69 | 129 | 198
  Week 144 | -73.1 (50.0) | -86.2 (57.8) | -81.6 (55.4)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | -66.1 (24.7) | -99.4 (48.3) | -86.1 (42.4)

4. Secondary Outcome: Absolute Change From Baseline in Calculated LDL-C (mmol/L) at Weeks 8, 24, 48, 72, 96, 120, 144 and 168
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, and 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
mmol/L
  Week 8: number analyzed (Participants) | 306 | 611 | 917
  Week 8 | -1.729 (1.180) | -1.738 (1.273) | -1.735 (1.242)
  Week 24: number analyzed (Participants) | 305 | 621 | 926
  Week 24 | -1.821 (1.282) | -1.883 (1.356) | -1.863 (1.332)
  Week 48: number analyzed (Participants) | 309 | 609 | 918
  Week 48 | -1.757 (1.286) | -1.914 (1.405) | -1.861 (1.368)
  Week 72: number analyzed (Participants) | 293 | 594 | 887
  Week 72 | -1.843 (1.154) | -1.940 (1.411) | -1.908 (1.332)
  Week 96: number analyzed (Participants) | 236 | 475 | 711
  Week 96 | -1.818 (1.190) | -1.965 (1.426) | -1.916 (1.353)
  Week 120: number analyzed (Participants) | 188 | 352 | 540
  Week 120 | -1.874 (1.180) | -1.949 (1.546) | -1.923 (1.428)
  Week 144: number analyzed (Participants) | 69 | 129 | 198
  Week 144 | -1.894 (1.294) | -2.232 (1.498) | -2.114 (1.436)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | -1.712 (0.641) | -2.574 (1.252) | -2.229 (1.098)

5. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) Over Time
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, and 168
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percentage of participants
  Baseline | 12.1 | 11.5 | 11.7
  Week 8: number analyzed (Participants) | 321 | 648 | 969
  Week 8 | 71.0 | 86.1 | 81.1
  Week 24: number analyzed (Participants) | 305 | 621 | 926
  Week 24 | 77.0 | 75.7 | 76.1
  Week 48: number analyzed (Participants) | 309 | 609 | 918
  Week 48 | 77.7 | 76.4 | 76.8
  Week 72: number analyzed (Participants) | 293 | 594 | 887
  Week 72 | 82.9 | 77.6 | 79.4
  Week 96: number analyzed (Participants) | 236 | 475 | 711
  Week 96 | 79.2 | 76.8 | 77.6
  Week 120: number analyzed (Participants) | 188 | 352 | 540
  Week 120 | 78.2 | 76.7 | 77.2
  Week 144: number analyzed (Participants) | 69 | 129 | 198
  Week 144 | 72.5 | 74.4 | 73.7
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | 75.0 | 83.3 | 80.0

6. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) Over Time
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, and 168
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percentage of participants
  Baseline | 0.9 | 1.2 | 1.1
  Week 8: number analyzed (Participants) | 321 | 648 | 969
  Week 8 | 47.4 | 66.4 | 60.1
  Week 24: number analyzed (Participants) | 305 | 621 | 926
  Week 24 | 53.4 | 53.1 | 53.2
  Week 48: number analyzed (Participants) | 309 | 609 | 918
  Week 48 | 51.1 | 53.5 | 52.7
  Week 72: number analyzed (Participants) | 293 | 594 | 887
  Week 72 | 57.0 | 53.2 | 54.5
  Week 96: number analyzed (Participants) | 236 | 475 | 711
  Week 96 | 53.0 | 56.4 | 55.3
  Week 120: number analyzed (Participants) | 188 | 352 | 540
  Week 120 | 52.7 | 50.9 | 51.5
  Week 144: number analyzed (Participants) | 69 | 129 | 198
  Week 144 | 46.4 | 48.1 | 47.5
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | 50.0 | 33.3 | 40.0

7. Secondary Outcome: Percentage of Participants With Calculated LDL-C <70 mg/dL (1.81mmol/L) and/or >=50% Reduction in Calculated LDL-C From Baseline (if Calculated LDL-C >=70 mg/dL [1.81mmol/L]) Over Time
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, and 168
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percentage of participants
  Baseline | 0.9 | 1.2 | 1.1
  Week 8: number analyzed (Participants) | 321 | 648 | 969
  Week 8 | 49.5 | 67.1 | 61.3
  Week 24: number analyzed (Participants) | 305 | 621 | 926
  Week 24 | 54.1 | 54.3 | 54.2
  Week 48: number analyzed (Participants) | 309 | 609 | 918
  Week 48 | 52.1 | 54.5 | 53.7
  Week 72: number analyzed (Participants) | 293 | 594 | 887
  Week 72 | 57.3 | 54.4 | 55.4
  Week 96: number analyzed (Participants) | 236 | 475 | 711
  Week 96 | 53.0 | 57.7 | 56.1
  Week 120: number analyzed (Participants) | 188 | 352 | 540
  Week 120 | 53.2 | 53.1 | 53.1
  Week 144: number analyzed (Participants) | 69 | 129 | 198
  Week 144 | 46.4 | 48.8 | 48.0
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | 50.0 | 33.3 | 40.0

8. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Weeks 8, 24, 48, 72, 96, 120, 144 and 168
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, and 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percent change
  Week 8: number analyzed (Participants) | 310 | 618 | 928
  Week 8 | -38.1 (24.8) | -37.6 (26.6) | -37.8 (26.0)
  Week 24: number analyzed (Participants) | 310 | 625 | 935
  Week 24 | -40.6 (25.5) | -40.4 (27.9) | -40.5 (27.1)
  Week 48: number analyzed (Participants) | 310 | 616 | 926
  Week 48 | -39.7 (25.5) | -40.6 (27.6) | -40.3 (26.9)
  Week 72: number analyzed (Participants) | 294 | 597 | 891
  Week 72 | -40.8 (22.6) | -40.3 (26.5) | -40.5 (25.3)
  Week 96: number analyzed (Participants) | 240 | 481 | 721
  Week 96 | -39.9 (23.5) | -40.5 (26.6) | -40.3 (25.6)
  Week 120: number analyzed (Participants) | 188 | 358 | 546
  Week 120 | -41.4 (22.1) | -38.4 (29.7) | -39.5 (27.3)
  Week 144: number analyzed (Participants) | 70 | 132 | 202
  Week 144 | -39.8 (22.9) | -41.8 (24.0) | -41.1 (23.6)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | -40.7 (12.3) | -47.7 (18.8) | -44.9 (16.1)

9. Secondary Outcome: Percent Change From Baseline in Total-cholesterol at Weeks 8, 24, 48, 72, 96, 120, 144 and 168
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, and 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percent change
  Week 8: number analyzed (Participants) | 310 | 618 | 928
  Week 8 | -27.9 (19.3) | -27.7 (20.7) | -27.7 (20.2)
  Week 24: number analyzed (Participants) | 310 | 625 | 935
  Week 24 | -30.1 (20.3) | -30.2 (21.6) | -30.1 (21.2)
  Week 48: number analyzed (Participants) | 310 | 616 | 926
  Week 48 | -29.0 (20.5) | -30.0 (21.6) | -29.7 (21.2)
  Week 72: number analyzed (Participants) | 294 | 597 | 891
  Week 72 | -29.9 (18.0) | -30.1 (20.8) | -30.0 (19.9)
  Week 96: number analyzed (Participants) | 240 | 481 | 721
  Week 96 | -28.9 (18.3) | -29.9 (21.1) | -29.6 (20.2)
  Week 120: number analyzed (Participants) | 188 | 358 | 546
  Week 120 | -30.2 (17.2) | -28.4 (22.8) | -29.0 (21.0)
  Week 144: number analyzed (Participants) | 70 | 132 | 202
  Week 144 | -29.1 (18.2) | -31.3 (19.1) | -30.5 (18.8)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | -32.3 (12.4) | -39.1 (14.3) | -36.4 (13.3)

10. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Weeks 8, 24, 48, 72, 96, 120, 144 and 168
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, and 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percent change
  Week 8: number analyzed (Participants) | 310 | 618 | 928
  Week 8 | 5.6 (17.1) | 6.6 (17.3) | 6.3 (17.3)
  Week 24: number analyzed (Participants) | 310 | 625 | 935
  Week 24 | 5.7 (17.4) | 5.8 (16.9) | 5.8 (17.1)
  Week 48: number analyzed (Participants) | 310 | 616 | 926
  Week 48 | 7.1 (17.8) | 7.2 (19.2) | 7.2 (18.7)
  Week 72: number analyzed (Participants) | 294 | 597 | 891
  Week 72 | 6.7 (17.6) | 7.2 (19.9) | 7.0 (19.1)
  Week 96: number analyzed (Participants) | 240 | 481 | 721
  Week 96 | 7.2 (18.8) | 7.2 (18.7) | 7.2 (18.7)
  Week 120: number analyzed (Participants) | 188 | 358 | 546
  Week 120 | 8.0 (18.4) | 8.1 (18.7) | 8.1 (18.6)
  Week 144: number analyzed (Participants) | 70 | 132 | 202
  Week 144 | 8.8 (19.2) | 8.8 (24.8) | 8.8 (23.0)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | -6.6 (26.2) | -0.3 (9.9) | -2.8 (17.1)

11. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides (TGs) at Weeks 8, 24, 48, 72, 96, 120, 144 and 168
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, and 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percent change
  Week 8: number analyzed (Participants) | 309 | 618 | 927
  Week 8 | 3.4 (40.5) | 3.5 (47.0) | 3.5 (44.9)
  Week 24: number analyzed (Participants) | 308 | 624 | 932
  Week 24 | 0.6 (39.9) | 1.0 (45.9) | 0.9 (44.0)
  Week 48: number analyzed (Participants) | 309 | 616 | 925
  Week 48 | 0.8 (37.5) | 5.1 (78.0) | 3.7 (67.2)
  Week 72: number analyzed (Participants) | 293 | 596 | 889
  Week 72 | 4.3 (43.3) | 3.6 (42.9) | 3.8 (43.0)
  Week 96: number analyzed (Participants) | 239 | 479 | 718
  Week 96 | 9.1 (53.2) | 9.3 (55.2) | 9.2 (54.5)
  Week 120: number analyzed (Participants) | 187 | 358 | 545
  Week 120 | -1.2 (35.3) | 10.8 (48.5) | 6.7 (44.8)
  Week 144: number analyzed (Participants) | 70 | 131 | 201
  Week 144 | 5.0 (38.0) | 7.7 (49.8) | 6.8 (45.9)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | -22.1 (21.9) | -10.3 (27.1) | -15.0 (24.6)

12. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Weeks 48, 96, 144 and 168
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 48, 96, 144, and 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percent change
  Week 48: number analyzed (Participants) | 307 | 606 | 913
  Week 48 | -15.0 (158.4) | -26.4 (40.2) | -22.6 (97.6)
  Week 96: number analyzed (Participants) | 239 | 474 | 713
  Week 96 | -13.9 (171.7) | -21.4 (132.7) | -18.9 (146.9)
  Week 144: number analyzed (Participants) | 69 | 129 | 198
  Week 144 | -20.1 (46.1) | -33.0 (25.0) | -28.5 (34.3)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | -30.3 (18.2) | -29.2 (15.4) | -29.6 (15.6)

13. Secondary Outcome: Percent Change From Baseline in Apolipoprotein-B (Apo-B) at Weeks 48, 96, 144, and 168
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 48, 96, 144, and 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percent change
  Week 48: number analyzed (Participants) | 308 | 607 | 915
  Week 48 | -36.9 (21.7) | -37.8 (23.4) | -37.5 (22.9)
  Week 96: number analyzed (Participants) | 238 | 475 | 713
  Week 96 | -36.9 (20.9) | -38.0 (22.9) | -37.6 (22.3)
  Week 144: number analyzed (Participants) | 69 | 129 | 198
  Week 144 | -33.9 (20.9) | -36.9 (21.3) | -35.9 (21.2)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | -38.0 (9.0) | -43.1 (20.7) | -41.1 (16.5)

14. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (Apo A-1) at Weeks 48, 96, 144, and 168
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 48, 96, 144, and 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
percent change
  Week 48: number analyzed (Participants) | 308 | 607 | 915
  Week 48 | 5.6 (14.5) | 5.8 (17.2) | 5.7 (16.3)
  Week 96: number analyzed (Participants) | 238 | 475 | 713
  Week 96 | 7.8 (15.4) | 8.5 (14.1) | 8.3 (14.5)
  Week 144: number analyzed (Participants) | 69 | 129 | 198
  Week 144 | 11.2 (16.3) | 10.2 (18.7) | 10.6 (17.8)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | 0.9 (19.3) | 3.9 (9.3) | 2.7 (13.2)

15. Secondary Outcome: Absolute Change From Baseline in Apo B/Apo A-1 Ratio at Weeks 48, 96, 144, and 168
Description: as for outcome 2
Time Frame: Parent Baseline, Weeks 48, 96, 144, and 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
Number analyzed (Participants) | 323 | 651 | 974
ratio
  Week 48: number analyzed (Participants) | 308 | 607 | 915
  Week 48 | -0.340 (0.245) | -0.361 (0.304) | -0.354 (0.286)
  Week 96: number analyzed (Participants) | 238 | 475 | 713
  Week 96 | -0.340 (0.228) | -0.375 (0.268) | -0.363 (0.256)
  Week 144: number analyzed (Participants) | 69 | 129 | 198
  Week 144 | -0.342 (0.242) | -0.414 (0.433) | -0.389 (0.379)
  Week 168: number analyzed (Participants) | 4 | 6 | 10
  Week 168 | -0.370 (0.161) | -0.498 (0.280) | -0.447 (0.238)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 176 post-treatment follow-up visit) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are treatment emergent that is AEs that developed/worsened and deaths that occurred during the 'on treatment' period (from the first dose of alirocumab in this study up to the last dose of alirocumab received in this study + 70 days).
Groups:
- Alirocumab to Alirocumab 75 or 150 mg Q2W: Alirocumab 75 mg or 150 mg SC injection Q2W added to stable LMT for up to 168 weeks in participants who received Alirocumab in the parent studies. Participants from parent study EFC12732 (NCT01617655) started with alirocumab 150 mg Q2W and participants from parent studies EFC12492 (NCT01623115), R727-CL-1112 (NCT01709500) and LTS11717 (NCT01507831) started with alirocumab 75 mg Q2W. Alirocumab doses could be either up-titrated from 75 to 150 mg Q2W or down-titrated from 150 to 75 mg Q2W from Week 12 or maintained according to the investigator judgement and LDL-C values.
- Alirocumab: All Participants: All participants who received alirocumab/placebo in the parent studies and received alirocumab 75 mg or 150 mg SC injection Q2W added to stable LMT for up to 168 weeks in this study.
Arm/Group | Placebo to Alirocumab 75 or 150 mg Q2W | Alirocumab to Alirocumab 75 or 150 mg Q2W | Alirocumab: All Participants
All-Cause Mortality (participants affected / at risk) | 4/330 | 7/655 | 11/985
Serious Adverse Events (participants affected / at risk) | 68/330 | 144/655 | 212/985
Other Adverse Events (participants affected / at risk) | 183/330 | 366/655 | 549/985
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to Alirocumab 75 or 150 mg Q2W (N=330) | Alirocumab to Alirocumab 75 or 150 mg Q2W (N=655) | Alirocumab: All Participants (N=985)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 6 | 8 | 14
Angina unstable (Cardiac disorders) | 4 | 5 | 9
Acute myocardial infarction (Cardiac disorders) | 2 | 4 | 6
Coronary artery disease (Cardiac disorders) | 2 | 4 | 6
Coronary artery stenosis (Cardiac disorders) | 3 | 3 | 6
Myocardial infarction (Cardiac disorders) | 2 | 3 | 5
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 4
Cardiac failure (Cardiac disorders) | 2 | 2 | 4
Cardiac failure congestive (Cardiac disorders) | 3 | 1 | 4
Ventricular tachycardia (Cardiac disorders) | 1 | 3 | 4
Aortic valve stenosis (Cardiac disorders) | 2 | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 2
Aortic valve disease (Cardiac disorders) | 1 | 0 | 1
Aortic valve disease mixed (Cardiac disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 1
Coronary artery thrombosis (Cardiac disorders) | 0 | 1 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 1
Mitral valve stenosis (Cardiac disorders) | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1
Hereditary non-polyposis colorectal cancer syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1
Glaucoma (Eye disorders) | 0 | 2 | 2
Optic ischaemic neuropathy (Eye disorders) | 1 | 1 | 2
Corneal decompensation (Eye disorders) | 1 | 0 | 1
Open angle glaucoma (Eye disorders) | 0 | 1 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 1
Retinal tear (Eye disorders) | 0 | 1 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 1 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Internal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 1
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 4 | 6
Chest pain (General disorders) | 1 | 2 | 3
Death (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 1 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1 | 1
Vascular stent occlusion (General disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 3 | 5
Cellulitis (Infections and infestations) | 0 | 3 | 3
Bronchitis (Infections and infestations) | 0 | 2 | 2
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Hepatitis E (Infections and infestations) | 0 | 2 | 2
Catheter site infection (Infections and infestations) | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 1
Corneal abscess (Infections and infestations) | 1 | 0 | 1
Cystitis bacterial (Infections and infestations) | 0 | 1 | 1
Device related sepsis (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 1 | 1
Peritoneal abscess (Infections and infestations) | 1 | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 1
Stitch abscess (Infections and infestations) | 1 | 0 | 1
Viral myocarditis (Infections and infestations) | 0 | 1 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Heart rate irregular (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 5 | 7
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Chronic lymphocytic leukaemia stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastatic glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 6 | 7
Transient ischaemic attack (Nervous system disorders) | 0 | 6 | 6
Amnesia (Nervous system disorders) | 2 | 0 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 2 | 2
Presyncope (Nervous system disorders) | 1 | 1 | 2
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 1
Dementia (Nervous system disorders) | 0 | 1 | 1
Embolic cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Focal dyscognitive seizures (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 1
Hemiplegia (Nervous system disorders) | 0 | 1 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1 | 1
Sensory loss (Nervous system disorders) | 0 | 1 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 1 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Device defective (Product Issues) | 0 | 1 | 1
Device loosening (Product Issues) | 0 | 1 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 1
Alcoholism (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Delirium tremens (Psychiatric disorders) | 1 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 4
Nephrolithiasis (Renal and urinary disorders) | 1 | 3 | 4
Renal colic (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 2
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 1
Vaginal dysplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 2
Neurogenic shock (Vascular disorders) | 1 | 1 | 2
Air embolism (Vascular disorders) | 0 | 1 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 1 | 1
Intermittent claudication (Vascular disorders) | 0 | 1 | 1
Malignant hypertension (Vascular disorders) | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to Alirocumab 75 or 150 mg Q2W (N=330) | Alirocumab to Alirocumab 75 or 150 mg Q2W (N=655) | Alirocumab: All Participants (N=985)
Diarrhoea (Gastrointestinal disorders) | 19 | 43 | 62
Influenza like illness (General disorders) | 12 | 40 | 52
Injection site reaction (General disorders) | 26 | 28 | 54
Bronchitis (Infections and infestations) | 19 | 41 | 60
Influenza (Infections and infestations) | 34 | 61 | 95
Upper respiratory tract infection (Infections and infestations) | 31 | 71 | 102
Urinary tract infection (Infections and infestations) | 21 | 28 | 49
Viral upper respiratory tract infection (Infections and infestations) | 51 | 93 | 144
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 53 | 87
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 56 | 82
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 44 | 59
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 31 | 49
Hypertension (Vascular disorders) | 13 | 37 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2015-07-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT01954394/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT01954394/SAP_001.pdf